CLINICAL TRIAL: NCT05760326
Title: Diagnostic and Prognostic Role of Clot Analysis in Stroke Patients
Acronym: DICAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5153
Record Dates: First submitted 2023-02-27; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-02

CONDITIONS: Stroke, Acute; Atherosclerosis; Atrial Fibrillation
MeSH Terms: conditions — Stroke; Atherosclerosis; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
BACKGROUND AND RATIONALE OF THE STUDY

The analysis of the composition of the clot constitutes a promising tool for investigating the possible pathogenetic mechanisms underlying ischemic stroke. This analysis was made possible thanks to the numerous mechanical thrombectomy operations which have now become routine.

Several studies have attempted to explore the possible relationship between the primary site of thrombus formation and clot composition, reporting that cardioembolic stroke may have a higher percentage of platelet-rich areas than noncardioembolic thrombosis. However, the data are conflicting and do not seem to support an association between clot histology and etiology. Furthermore, thrombus composition appears to influence thrombolysis and the efficacy of thrombectomy. For example, fibrin-rich thrombi appear to reduce the effectiveness of thrombolytic treatment and require more steps with mechanical thrombectomy treatment.

Primary ENDPOINT:

Evaluate how clot composition relates to stroke etiology according to the TOAST classification.

Secondary ENDPOINT:

* relationship between different clot components and the degree of thrombectomy recanalization as defined by treatment modified cerebral ischemia score (mTICI).
* relationship between the different components of the clot and the number of steps required to achieve recanalization.
* relationship between the different clot components and outcome indicators (NIHSS score and mRS score).

TARGET POPULATION Patients with ischemic stroke with occlusion of large intracranial vessels will be included in the study if deemed suitable for mechanical thrombectomy therapy in accordance with national and international guidelines.

INCLUSION CRITERIA

* age > 18 years;
* Patients diagnosed with large vessel occlusion stroke in the emergency room CT Angio-study, undergoing mechanical thrombectomy procedure.
* Recovered thrombus available for analysis

EXCLUSION CRITERIA

● Lack of written informed consent.

MATERIALS AND METHODS The clot will be portioned. Part of the sample will be fixed in a 10% formalin solution (3.7% formaldehyde), part will be frozen in liquid nitrogen. Within 24-48 hours of fixation, formalin-fixed thrombi will be dehydrated by increasing the concentration of ethanol (70%, -80%, -95%, 100%) and paraffin-embedded allowing good preservation of tissue morphology and easy long-term storage. The included samples will be sectioned along the major axis of the thrombus, in slices with a thickness between 4 and 5 µm.

Base staining will be used to visualize RBC, PLT and fibrin.

* Hematoxylin and Eosin (H&E) will allow visualization of general thrombus structures and identification of aggregates of fibrin/platelets (colored pink), red blood cells (red), and nucleated cells (dark blue).
* Martius Scarlet Blue (MSB), selectively stains fibrin (dark pink/red), red blood cells (yellow) and collagen (blue
* Mallory-Azan for collagen and phosphotungstic acid hematoxylin for fibrin.
* immunohistochemistry to detect the presence of

  * Platelets (CD42-Gp-Ib+, CD41a-Gp-IIb/IIIa+, CD61-GpIIIa),
  * white blood cells (CD45+, common leukocyte antigen), or monocytes/macrophages (CD14+, CD1a+, CD68+),
  * T lymphocytes (CD3+, CD8/CD4+), or natural killers (CD16+, CD56+), or mobile premature endothelial cells and blood progenitors (CD34+), or neutrophils (CD45+, CD16+), or fibrinogen or von Willebrand factor.

DETAILED DESCRIPTION:
2. BACKGROUND

Stroke is the second leading cause of death and the third cause of disability worldwide. The majority of strokes are ischemic, mainly caused by blood thrombi occluding a cerebral vessel1. According to the TOAST classification2, four cause of stroke due to large vessel occlusion (LVO) can be identified: atherosclerosis, cardioembolic, other determined etiology (like dissection) or other undetermined causes. Strokes without a defined etiology are now called "embolic stroke of undetermined nature" (ESUS)3. This definition implies the presence of an undefined embolic source as the cause of the stroke. Not knowing the origin of the embolus, the best medical therapy in these patients is actually matter of debate4-6. Research on this topic is focusing on finding a laboratory or radiologic marker capable of clearly identified the embolic source and guide in the choice of the best medical therapy7,8.

Revascularization strategy, such as thrombolysis and thrombectomy, represent the gold standard therapy during stroke acute phase, in particular for patients with large vessel occlusion (LVO). From 2015 a growing body of evidence showed the efficacy of endovascular procedures in stroke patients and, furthermore, allowed for the first time the opportunity to collect thrombus material for research purposes9,10.

3. OBJECTIVES

The objective of this study is to evaluate how clot composition is related to stroke etiology according to the TOAST classification. Furthermore, we will also study the relationship between different clot components and thrombectomy grade of recanalization as defined by the modified treatment in cerebral ischemia score (mTICI) and the number of required passes to achieve recanalization.

4. STUDY DESIGN Study population

Patients hospitalized in the - Catholic University of the Sacred Heart, Policlinico Gemelli - Catholic University - Rome, with a stroke due to LVO treated with mechanical thrombectomy will be presented the study.

Patient will be enrolled upon their presentation to the emergency department. The usual clinical practice will be followed.

Considering the emergency setting and the impossibility for most patients to provide a valid and informed consent before e immediately after the procedures, retrieved thrombi will be collected but not analyze. An informed consent to the study will be collect in the following day. Should the patient refuse the participation, the thrombus will be discarded and the patient will be considered as a drop out from the study.

Investigators plan to include 30 patients with acute ischemic stroke due to LVO treated with mechanical thrombectomy.

Patient's characteristics Ischemic stroke patients with LVO will be included in the study if considered suitable for mechanical thrombectomy therapy in accordance with national and international guidelines.

Inclusion criteria

* age > 18 years;
* Patients with a diagnosis of large vessel occlusion stroke at the Angio-CT study performed in the ER, undergoing a mechanical thrombectomy procedure.
* Thrombus retrieved available for analysis

Exclusion criteria:

* Deny informed consent

  5. ENDPOINTS Primary endpoint
* To evaluate the association between thrombus composition, studied through histological and immunohistochemical coloration, and stroke etiology according to the TOAST classification. In particular, TOAST voices for etiological category will be dichotomize between "cardioembolic" and "not cardioembolic" (the latter including "large vessel occlusion", "other determined etiologies" and "other undetermined etiologies").

Secondary endpoints

* To evaluate the association between thrombus composition and mechanical thrombectomy outcome.
* To evaluate the association between thrombus composition and number of passes needed to obtain recanalization.

"Correlation" endpoints

• To evaluate the correlation between thrombus composition and global outcome variable such as the National Institutes of Health Stroke Scale (NIHSS) at seven days and nineteen days after the event and the modified ranking scale (mRS) at three months.

6. METHODS AND ASSESSMENT

Clinical variables and neuroimaging studies The following data will be collected: medical history recording, demographic data (age, sex), potential vascular risk factors, (hypertension, diabetes mellitus, dyslipidemia, smoking, prior stroke/ transient ischemic attack (TIA), previous vascular diseases, previous antiplatelet treatment, congestive heart failure, hypertension, vascular disease, abnormal renal/liver function, bleeding history or predisposition, labile international normalized ratio, drugs/alcohol concomitantly), diagnosis of atrial fibrillation, Oxfordshire Community Stroke Project (OCSP) classification, previous treatment with thrombolysis, ASPECTS/pc-ASPECTS (based on TC scan performed 24 h after acute stroke), andHemorrhagic trasformation subtype. At three months follow-up, the following data will be collected: intracranial bleeding, major and minor bleeding, blood transfusion, hospitalization, deaths, modified Rankin Scale (mRS) score, adherence to treatment, stroke recurrence, and myocardial infarction. Laboratory tests, blood counts, biochemistry and coagulation tests, 12-lead ECG, chest radiography, carotid ultrasonography and Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) will be performed at admission and during the hospitalization.

To evaluate neurologic deficit, the National Institute of Health Stroke Scale (NIHSS) will be performed at admission, 24, 48, 72 h, 7 days and/or at discharge, and at 3 months.

Functional outcome will be evaluated at discharge and at 3 months by modified rankin scale (mRS). Stroke etiology will be classified according to TOAST criteria for ischemic stroke. TOAST voices for etiological category will be dichotomize between "cardioembolic" and "not cardioembolic" (the latter including "large vessel occlusion", "other determined etiologies" and "other undetermined etiologies").

To evaluate infarct volume, and control hemorrhagic evolution a CT will be performed between 24 ours from treatment. Infarct volume will be quantified in cubic centimeters (cm3) and assessed according to the formula 0.5xAxBxC, where A direction and C to the number of 10mm slices where infarct volume is present [20]. All neuroimaging evaluations will be made by the a neuroradiologist blinded to clinical and laboratory data.

Specimen fixation and sectioning Retrieved thrombi will be portioned. Part of the specimen will be fixed in a solution of 10% formalin (3,7% formaldehyde), part will be frozen in liquid azote. Within 24-48 hours from fixation, formalin-fixed thrombi will be dehydrated via increasing concentration of ethanol (70%, -80%, -95%, 100%) and embedded in paraffin allowing a good preservation of tissue morphology and easy long-term storage. Included samples will be sectioned along the major axis of the thrombus, in slice with a 4 to 5 µm of thickness.

Staining Base coloration will be employed to visualize RBC, PLT and fibrin. Hematoxylin and eosin staining (H&E) will allow to visualize the general overall structures of the thrombus and the identification of fibrin/platelet aggregates (colored in pink), RBC (red) and nucleated cells (dark blue). The Martius Scarlet Blue (MSB) staining, instead, will selectively stain fibrin (Dark pink/red), RBC (yellow) and collagen (Blue). RBC-rich fibrin-poor material will appears red on H&E staining and yellow on MSB, while RBC-poor/fibrin-rich areas will appear as light pink areas on H&E staining and pink to red areas on MSB. Since platelets are only present in large amount in RBC-poor fibrin-rich areas, thrombi will be divided in: RBC-rich/Platelets-poor, mixed and platelets-rich/RBC-poor. Additional base coloration will include Mallory-Azan for collagen and phosphotungstic acid hematoxylin for fibrin. Furthermore, immunohistochemical staining will be employed to detect the presence of Platelets (CD42-Gp-Ib+, CD41a-Gp-IIb/IIIa+, CD61-GpIIIa), white blood cells (CD45+, leukocyte common antigen), monocyte/macrophages (CD14+, CD1a+, CD68+), T lymphocytes (CD3+, CD8/CD4+), Natural Killer cells (CD16+, CD56+), premature endothelial and blood progenitor cells (CD34+), Neutrophils (CD45+, CD16+), Fibrinogen and Von Willebrand factor.

Analysis Standardized quantification algorithms to calculate thrombus composition will be employed. Computational color-based segmentation analysis by the means of ImageJ (Rasband, W.S., ImageJ, U. S. National Institutes of Health, Bethesda, Maryland, USA, https://imagej.nih.gov/ij/, 1997-2018.) will allow to apply thresholds for color and thus selective quantification of specific colors/components, providing data in automated manner about the percentage of total thrombus areas.

7. STATISTICAL ANALYSIS

In this study 28 consecutive patients fulfilling selection criteria will be included. According to the analysis of Kim (2015) strong differences in mean percentages in clot composition between the two subgroups are reported, therefore it is possible to make an hypothesis of an effect size equal to or greater than 1; using the Student's t-test this sample size of 28 patients (increased to 30 for possible technical difficulties) included in one of the two groups determined by the TOAST classification will have a power of 80% to detect such differences at a significance level of 5% (two-tailed). Statistical analyses will be performed using the IBM-SPSS, Statistical Package for Social Science (SPSS) v.20. Kolmogorov-Smirnov test will be used to evaluate data distribution: in case of deviation from normality U test di Mann-Whitney or Kruskal-Wallis test will be used for comparisons among two or more groups; in case of respect of normality assumptions Students' t-test or analysis of variance will be considered. Association between dichotomomic items will be evaluated using the Fisher exact test or χ2, as appropriate. Due to the explorative approach of this study no adjustment will be made for multiple testing.

8. ETHICAL PRINCIPLES

This study will be conducted in accordance with the principles laid down by the 18th World Medical Assembly (Helsinki, 1964) and all applicable amendments laid down by the World Medical Assemblies, and the ICH guidelines for good clinical practice (GCP).

9. INFORMED CONSENT

The Investigator should fully inform the patient of all pertinent aspects of the study including the written information giving approval/favorable opinion by the Ethics Committee (IRB/IEC). All participants should be informed to the fullest extent possible about the study, in language and terms they are able to understand.

Prior to thrombus analysis, the written informed consent form should be signed, name filled in and personally dated by the patient or by the patient's legally acceptable representative, and by the person who conducted the informed consent discussion. A copy of the signed and dated written informed consent form will be provided to the patient.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years;
* Patients with a diagnosis of large vessel occlusion stroke at the Angio-CT study performed in the ER, undergoing a mechanical thrombectomy procedure.
* Thrombus retrieved available for analysis

Exclusion Criteria:

• Deny informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in the - Catholic University of the Sacred Heart, Policlinico Gemelli - Catholic University - Rome, with a stroke due to LVO treated with mechanical thrombectomy will be presented the study.
  Patient will be enrolled upon their presentation to the emergency department. The usual clinical practice will be followed.
  Considering the emergency setting and the impossibility for most patients to provide a valid and informed consent before e immediately after the procedures, retrieved thrombi will be collected but not analyze. An informed consent to the study will be collect in the following day. Should the patient refuse the participation, the thrombus will be discarded and the patient will be considered as a drop out from the study.
  Investigators plan to include 30 patients with acute ischemic stroke due to LVO treated with mechanical thrombectomy.
Sampling Method: Probability Sample
Enrollment: 13 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Clot - TOAST correlation | 1 year
  • To evaluate the association between thrombus composition, studied through histological and immunohistochemical coloration, and stroke etiology according to the TOAST classification. In particular, TOAST voices for etiological category will be dichotomize between "cardioembolic" and "not cardioembolic" (the latter including "large vessel occlusion", "other determined etiologies" and "other undetermined etiologies").

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli, IRCCS, Rome, Italy